CLINICAL TRIAL: NCT06086730
Title: Comparison Of Blow Bottle Positive Expiratory Pressure (BBPEP) Versus Acapella on Oxygenation ,Peak Expiratory Flow Rate (PEFR) Among Patient With Chronic Bronchitis
Brief Title: Comparison Of Blow Bottle Positive Expiratory Pressure (BBPEP) Versus Acapella Among Patient With Chronic Bronchitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/0347
Record Dates: First submitted 2023-10-11; First posted 2023-10-17 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Chronic Bronchitis
Keywords: alveolar collapse,hypersecreation,airway obstruction
MeSH Terms: conditions — Bronchitis, Chronic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- blow bottle positive expiratory pressure (Experimental): Water was poured into a 1 L plastic container until it reached a 10 cm height. A 30 cm long tube was put into the water in the bottle, 8 cm deep. The participants were instructed to close their mouths around the tubing in the apparatus for three seconds to produce bubbles, do this for a total of 10 breaths, perform two huffs, then cough. Such exhalations were conducted in two sets of ten, with a five-minute pause in between. For each subject, a fresh, disposable tube and bottle were utilized
  Interventions: Device: blow bottle positive expiratory pressure
- acapella (Active Comparator): Make sure the frequency adjustment dial has been rotated counterclockwise to the lowest frequency-resistance setting before using the Acapella for the first time. On a chair, adopt a straight stance. maintaining a straight back and relaxing your elbows on a table. Now gradually tilt your head upward to maintain the opening of your upper airways. Inhale more deeply than you frequently do. Make sure your lips are encircling the mouthpiece, then blow into the device with a strong expiration. You should ideally blow out roughly twice as quickly as usual. For around ten breaths. Make careful to expel to clear the secretions from the airways after the final try. You can even conduct 2 to 3 "huffs" to improve secretion elimination when necessary. It should be noted that while using the device, you must be capable of exhale for a minimum of three to four seconds.
  Interventions: Device: acapella

INTERVENTIONS:
Device: blow bottle positive expiratory pressure — Water was poured into a 1 L plastic container until it reached a 10 cm height. A 30 cm long tube was put into the water in the bottle, 8 cm deep. The participants were instructed to close their mouths around the tubing in the apparatus for three seconds to produce bubbles, do this for a total of 10 breaths, perform two huffs, then cough. Such exhalations were conducted in two sets of ten, with a five-minute pause in between. For each subject, a fresh, disposable tube and bottle were utilized,Because it is a homemade device and can be used with less equipment and with more ease at home . patient perform session three day per week for the duration of 8 weeks , each session last for 35-40 minutes.
  Arms: blow bottle positive expiratory pressure
Device: acapella — Make sure the frequency adjustment dial has been rotated counterclockwise to the lowest frequency-resistance setting before using the Acapella for the first time.On a chair, adopt a straight stance. maintaining a straight back and relaxing your elbows on a table. Now gradually tilt your head upward to maintain the opening of your upper airways.Inhale more deeply than you frequently do. Make sure your lips are encircling the mouthpiece, then blow into the device with a strong expiration.You should ideally blow out roughly twice as quickly as usual.For around ten breaths, keep going like this.Make careful to expel to clear the secretions from the airways after the final try. You can even conduct 2 to 3 "huffs" to improve secretion elimination when necessary.It should be noted that while using the device, you must be capable of exhale for a minimum of three to four seconds. patient perform session three day per week for the duration of 8 weeks , each session last for 35-40 minutes
  Arms: acapella

SUMMARY:
Comparison of Blow Bottle Positive Expiratory pressure(BBPEP)versus acapella on Oxygenation ,peak Expiratory Flow Rate(PEFR)among patient with chronic bronchitis.

DETAILED DESCRIPTION:
Worldwide most of the people belong to all age group may affected with Non communicable diseases(NCD) which leads them toward death globally . According to stats World Health Organization (WHO) declares about 41 million people are died due to NCD which means about 71 %people are died globally due to this .Chronic Respiratory diseases are one of the main non communicable disease . About 9.0 million(3.6%) adult belong to age group of 18 or older may suffer from chronic bronchitis . Hallmark of chronic bronchitis is that cough and sputum production for more than >3months in each of at least two connective years. Chronic bronchitis effects every third person having COPD but it may effect any body who had normal pulmonary functions. Now a days positive expiratory pressure (PEP)devices are used along Cardio Pulmonary Therapy(CPT) .PEP devices are help full in mobilize the secretion in lower respiratory tract , may also beneficial in collateral ventilation ,mucous secretion and most importantly optimize functional residual capacity among people who had pulmonary complications. Many PEP devices are available in market but BBPEP is in low cost and are easily in approach of every single person .PEP is non invasive technique used to improve clinical outcome .

In this study investigator compare the effect of BBPEP and Acapella in participant having chronic bronchitis .In case of BBPEP patient expires against resistance of water column which increase PEP ( positive expiratory pressure ) in inlet which transferred airway patients lungs this will keep the alveoli patent or may recruit the collapsed alveoli. This will decrease airway resistance and improve lung compliance . As airway resistance decreases the amount of SPO2 AND PEFR also improved . participant are randomly assigned into two different group GROUP(A) AND GROUP(B) Group (A) receive intervention by using BBPEP device along with deep breathing exercises group (B)participant use acapella devices so out come will be measured participant rotate the device toward positive(+) sign to increase resistance or may rotate device to minus (-) to decrease resistance participant is in comfortable short sitting position ask him to take deep breath and hold it for 3 sec nose clip attached to the participant participant lips sealed mouthpiece ask him to exhale into mouth piece maneuver repeated for 10 to 12 breath with 3 to 4 huffs all the steps repeated for 15 minute. study will be carried out for 8 weeks , 3 days per week. Outcome variables will be Peak flow meter , pulse oximeter ,casa q scale ,heart rate, respiratory rate blood pressure. Data will be analyzed on SPSS-25.

ELIGIBILITY:
Inclusion Criteria

* Participant having chronic bronchitis both male and female.
* Presence of chronic bronchitis I-e daily cough and sputum production for at least 3 months each year during the past 2 years.
* Current smoker or ex smoker with 5 packs years of smoking history.
* Participant willing to participate.
* Presence of air flow obstruction by spirometry(GOLD stage 2).
* Participant with stable hemodynamic .

Exclusion Criteria:

* History of cough syncope.
* participant who required intubation.
* Participant who is critically ill.
* Participant who required functional dependency.
* Participant having angina at rest or in minor effort.
* Participant having cardiac arrhythmia.
* Participant having severe airway obstruction I-e GOLD stage 4
* Participant with hemodynamic instability having heart rate >120 bpm.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
pulse oximeter | 8 weeks
  Pulse oximeter that measures the proportion of oxygenated hemoglobin in the blood in pulsating vessels, especially the capillaries of the finger or ear.
peak expiratory flow rate (PEFR) | 8 weeks
  Peak expiratory flow rate is the volume of air expelled from the lungs in one quick exhalation and is reliable indicator of ventillation adequacy as well as air flow obstruction .The normal peak flow value can range from person to person and is dependent upon factors such as sex ,age height
casa q scale | 8 weeks
  The cough and sputum assessment questionnaire (CASA-Q) was used to measure the severity and impact of cough and sputum in patients with COPD and chronic bronchitis. CASA-Q scores of each domain demonstrated significant association with HRQoL impairment CASA-Q was strongly lower when chronic bronchitis was present, but multivariate analyses demonstrated that the association of HRQoL impairment was greater with the cough impact domain score than with the usual definition of chronic bronchitis. The CASA-Q targets cough and sputum by an original approach assessing both the symptoms and impacts in dailyactivities within the last 7 days. Each item is answered ranging from never to always or from not at all to a lot / extremely as applicable each type is answered using five categories.

CONTACTS AND LOCATIONS:
Overall Officials: Sumera abdulhameed, MS, Principal Investigator — Riphah International University
Locations (1):
- Govt .Mian Meer Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liverani B, Nava S, Polastri M. An integrative review on the positive expiratory pressure (PEP)-bottle therapy for patients with pulmonary diseases. Physiother Res Int. 2020 Jan;25(1):e1823. doi: 10.1002/pri.1823. Epub 2019 Nov 25. PMID 31762162
- [Background] Widysanto A, Goldin J, Mathew G. Chronic Bronchitis. 2025 Feb 6. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK482437/ PMID 29494044
- [Background] Kim V, Criner GJ. Chronic bronchitis and chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2013 Feb 1;187(3):228-37. doi: 10.1164/rccm.201210-1843CI. Epub 2012 Nov 29. PMID 23204254
- [Background] Sehlin M, Ohberg F, Johansson G, Winso O. Physiological responses to positive expiratory pressure breathing: a comparison of the PEP bottle and the PEP mask. Respir Care. 2007 Aug;52(8):1000-5. PMID 17650355
- [Background] Patterson JE, Hewitt O, Kent L, Bradbury I, Elborn JS, Bradley JM. Acapella versus 'usual airway clearance' during acute exacerbation in bronchiectasis: a randomized crossover trial. Chron Respir Dis. 2007;4(2):67-74. doi: 10.1177/1479972306075483. PMID 17621572
- [Background] Sharma P, Prem V, Jain S. Immediate Effects of Acapella(R) on Dynamic Lung Compliance in Mechanically Ventilated Patients with Acute Respiratory Distress Syndrome: A Case Series. Indian J Crit Care Med. 2018 Feb;22(2):100-102. doi: 10.4103/ijccm.IJCCM_157_17. PMID 29531450